CLINICAL TRIAL: NCT05839496
Title: Effects of Cervical Stabilization Training on Individuals With Headache
Brief Title: Cervical Stabilization Training on Individuals With Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Clinical associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 730
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Headache
Keywords: Headache; Neck pain; Exercise
MeSH Terms: conditions — Headache; Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical Stabilization Training Group (Experimental): The Cervical Stabilization Training Group applied cervical stabilization training three times a week for 8 weeks. Each session was completed in 45 minutes.
  Interventions: Other: Cervical stabilization exercises
- Control Group (No Intervention): Control Group continued their medical treatment and they did not participate in any treatment for eight weeks.

INTERVENTIONS:
Other: Cervical stabilization exercises — Patients learned the activation of deep cervical flexor and extensor muscles. Then, during the activity of deep cervical muscles, superficial cervical muscles and upper extremity muscles were also strengthened. Thus, it was aimed to strengthen all neck muscles and upper extremity muscles in different positions synchronously and to increase their endurance.
  Arms: Cervical Stabilization Training Group

SUMMARY:
Headache is a common health problem. The most common headaches worldwide are migraine, tension-type headache (TTH), and cervicogenic headache (CGH). Due to the close anatomical relationship between the head and the cervical region, neck pain accompanies these headaches. The effects of cervical stabilization training including all of the cervical regions, thoracic regions, and the upper extremities in individuals with headaches are not yet known.

DETAILED DESCRIPTION:
Headache is a common health problem. The most common headaches worldwide are migraine, tension-type headache (TTH), and cervicogenic headache (CGH). Due to the close anatomical relationship between the head and the cervical region, neck pain accompanies these headaches. Most of the previous studies examined the effects of exercise programs such as Cranio-Cervical Flexion Exercises (CCFE), posture exercises, muscle strengthening, and stretching exercises of the neck and shoulder on headaches. These studies presented the beneficial effects of CCFE which mostly targeted strengthening the superficial neck and shoulder muscles. However, the effects of cervical stabilization training including all of the cervical regions, thoracic regions, and the upper extremities in individuals with headaches are not yet known.

ELIGIBILITY:
Inclusion Criteria:

1. a clinical diagnosis of migraine, tension-type headache (TTH), and cervicogenic headache (CGH)
2. age between 18 and 55 years
3. being female
4. frequency of headaches at least once a week or more in the last year

Exclusion Criteria:

1. having a neurological and orthopedic disease such as Parkinson's, stroke, cognitive disorders, and temporomandibular joint dysfunction,
2. having any contraindication for exercise,
3. having any serious head and/or neck trauma,
4. being with menopause,
5. being included in a physiotherapy program for head and neck pain in the last 12 months.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity assessed by the VAS | Eight weeks
  The average headache severity and neck pain severity in the last month was also assessed by using the Visual Analogue Scale (VAS). A Visual Analogue Scale (VAS) is one of the pain rating scales. A VAS consists of a line, often 10 cm long, with verbal anchors at either end (e.g., "no pain" on the far left and "the most intense pain imaginable" on the far right). The patient places a mark at a point on the line corresponding to the patient's rating of pain intensity.
Forward head posture assessed by the craniovertebral angle | Eight weeks
  To evaluate the cervical posture, pictures were taken from the side to objectively measure the forward head posture. Patients were asked to stand straight and then relax while the camera was placed at shoulder level. After printing the pictures, the craniovertebral angle was measured to represent the degree of forward head posture. This angle was calculated by measuring the angle between a horizontal line drawn through the 7th cervical vertebra and a line connecting the tragus of the ear and C7 spinous process.
Deep cervical flexor muscles strength assessed by the stabilizer pressure biofeedback | Eight weeks
  Cranio-Cervical Flexion Test : To begin the test, the patient is lying on a table in a supine position with their neck in a neutral position. A biofeedback stabilizer device is then placed under the patient's neck to rest against the occiput and inflated to a baseline pressure of 20 mmHg. During the test, the patient is asked to close their mouth with a slight gap between their jaws and place their tongue on the upper palate. They are then instructed to nod their head as if saying "yes." In the first stage of the test, the patient is asked to increase the pressure by 2 mmHg and maintain this position at 22 mmHg for 10 seconds. The patient is then asked to relax. In subsequent stages of the test, the pressure is reset to the initial pressure of 20 mmHg, and the patient is asked to perform the same head movement for 10 repetitions to create a pressure of 4, 6, 8, and 10 mmHg, respectively, and maintain the pressure for 10 seconds in each movement.
Endurance of cervical muscles assessed by the chronometer | Eight weeks
  During the endurance test of cervical flexors, the patient is lying supıne position with the therapist's hand placed under their head. They are then asked to bring their chin closer to their chest, lifting their head about 2.5 cm and holding that position. The time they are able to maintain the position is recorded in seconds.
  During the endurance test of cervical extensors, the patient is lying down with their heads bent downwards and their heads and chest hanging over the bed, with a 2-kg sandbag placed on the back of their necks. They are then asked to lift their heads to a neutral position and hold their position. The time they are able to maintain the position is recorded in seconds.
Cervical joint range of motion assessed by the cervical range of motion instrument | Eight weeks
  The cervical joint range of motion was evaluated with a cervical joint range of motion measuring device. Active range of motion was measured in cervical flexion, extension, right rotation, left rotation, right lateral flexion, and left lateral flexion. Joint range of motion measurements were measured while the patient was sitting normally in an armless chair with a backrest.

SECONDARY OUTCOMES:
Disability level (headache) assessed by migraine disability rating scale | Eight weeks
  Migraine Disability Rating Scale: The Migraine Disability Assessment (MIDAS) questionnaire is a tool used to measure the impact of migraines on a person's daily life. It is a self-reported measure that assesses how much a person's headaches have affected their ability to perform daily activities, such as work, household chores, or social activities, over the past three months. The MIDAS questionnaire consists of five questions, with scores ranging from 0 to 270, and a higher score indicating a greater impact of migraine on daily activities.
  The Migraine Disability Rating Scale (MIDAS) can be used to classify the severity of a person's migraines into one of four categories:
  Grade I: Little or no disability, with a MIDAS score of 0-5. Grade II: Mild to moderate disability, with a MIDAS score of 6-10. Grade III: Moderate to severe disability, with a MIDAS score of 11-20. Grade IV: Severe disability, with a MIDAS score of more than 20.
Disability level (neck pain) assessed by the neck disability index | Eight weeks
  The Neck Disability Index (NDI): is a questionnaire that assesses the level of disability experienced by a person with neck pain. It was developed to measure the impact of neck pain on a person's ability to perform daily activities and to provide a standardized way of assessing disability due to neck pain. The NDI consists of 10 questions, each addressing a different aspect of daily life. The questions cover areas such as pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. The patient rates their level of disability for each question on a scale of 0 to 5, with 0 indicating no disability and 5 indicating complete disability. The scores for each question are then totaled. The maximum score is 50. The obtained score can be multiplied by 2 to produce a percentage score. Scoring intervals for interpretation, as follows:
  0 - 4 = no disability 5 - 14 = mild 15 - 24 = moderate 25 - 34 = severe above 34 = complete.
Health-related quality of life assessed by the short form 36 quality of life scale | Eight weeks
  The Short Form 36 Quality of Life Scale (SF-36): is a self-reported questionnaire used to assess an individual's overall health-related quality of life. It includes 36 questions and covers eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. To score the SF-36, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Higher scores indicate better health status and a mean score of 50 has been articulated as a normative value for all scales.
Sleep quality assessed by the Pittsburgh sleep quality index | Eight weeks
  The Pittsburgh Sleep Quality Index (PSQI): is a self-reported questionnaire that assesses an individual's sleep quality and disturbances over a one-month time period. The questionnaire consists of 19 questions that are grouped into seven categories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each category is scored on a scale of 0 to 3, with 3 indicating the greatest sleep disturbance. The seven category scores are then summed to produce a global PSQI score, which ranges from 0 to 21. A score of 5 or greater indicates poor sleep quality, while a score of 8 or greater is considered a severe sleep disturbance. The PSQI has been used in research studies and clinical settings to evaluate sleep quality and to identify individuals who may benefit from interventions to improve their sleep.
Mood assessed by the Beck depression inventory | Eight weeks
  The Beck Depression Inventory (BDI): is a self-report questionnaire that measures the severity of depression in individuals. The BDI consists of 21 questions or items, each of which has four possible responses. The questions cover a range of symptoms commonly associated with depression, such as sadness, loss of interest in activities, feelings of worthlessness or guilt, changes in appetite or sleep, and thoughts of self-harm. The responses are scored on a scale from 0 to 3, with higher scores indicating more severe depression. The total score ranges from 0 to 63, with scores of 0-9 indicating minimal depression, scores of 10-18 indicating mild depression, scores of 19-29 indicating moderate depression, and scores of 30 or higher indicating severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Guclu-Gunduz, Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-de-Las-Penas C, Florencio LL, Plaza-Manzano G, Arias-Buria JL. Clinical Reasoning Behind Non-Pharmacological Interventions for the Management of Headaches: A Narrative Literature Review. Int J Environ Res Public Health. 2020 Jun 9;17(11):4126. doi: 10.3390/ijerph17114126. PMID 32527071
- [Background] Castien R, De Hertogh W. A Neuroscience Perspective of Physical Treatment of Headache and Neck Pain. Front Neurol. 2019 Mar 26;10:276. doi: 10.3389/fneur.2019.00276. eCollection 2019. PMID 30972008
- [Background] Ashina S, Bendtsen L, Lyngberg AC, Lipton RB, Hajiyeva N, Jensen R. Prevalence of neck pain in migraine and tension-type headache: a population study. Cephalalgia. 2015 Mar;35(3):211-9. doi: 10.1177/0333102414535110. Epub 2014 May 22. PMID 24853166
- [Background] Edmondston SJ, Wallumrod ME, Macleid F, Kvamme LS, Joebges S, Brabham GC. Reliability of isometric muscle endurance tests in subjects with postural neck pain. J Manipulative Physiol Ther. 2008 Jun;31(5):348-54. doi: 10.1016/j.jmpt.2008.04.010. PMID 18558277
- [Background] Luedtke K, Basener A, Bedei S, Castien R, Chaibi A, Falla D, Fernandez-de-Las-Penas C, Gustafsson M, Hall T, Jull G, Kropp P, Madsen BK, Schaefer B, Seng E, Steen C, Tuchin P, von Piekartz H, Wollesen B. Outcome measures for assessing the effectiveness of non-pharmacological interventions in frequent episodic or chronic migraine: a Delphi study. BMJ Open. 2020 Feb 12;10(2):e029855. doi: 10.1136/bmjopen-2019-029855. PMID 32051295